CLINICAL TRIAL: NCT01913977
Title: Clinical Study to Determine the Optimal Operation Parameters During CO2 Removal With the Abylcap® System.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013/386
Record Dates: First submitted 2013-06-06; First posted 2013-08-01 (Estimated); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: ARDS (Acute Respiratory Distress Syndrome); Respiratory Acidosis
MeSH Terms: conditions — Acute Lung Injury; Acidosis, Respiratory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with mechanical ventilation (Experimental): Abylcap system with the oxygenator Lilliput2 as CO2 remover (Bellco, Italy).
  Interventions: Device: Abylcap® System: blood flow (QB): 200mL/min; gas flow (QG):7L/min; Device: Abylcap® System: blood flow (QB): 300mL/min; gas flow (QG):7L/min; Device: Abylcap® System: blood flow (QB): 400mL/min; gas flow (QG):7L/min; Device: Abylcap® System: blood flow (QB): 400mL/min; gas flow (QG):1.5L/min; Device: Abylcap® System: blood flow (QB): 400mL/min; gas flow (QG):3L/min; Device: Abylcap® System: blood flow (QB): 400mL/min; gas flow (QG):6L/min; Device: Abylcap® System: blood flow (QB): 400mL/min; gas flow (QG):8L/min

INTERVENTIONS:
Device: Abylcap® System: blood flow (QB): 200mL/min; gas flow (QG):7L/min — Abylcap settings
Device: Abylcap® System: blood flow (QB): 300mL/min; gas flow (QG):7L/min — Abylcap settings
Device: Abylcap® System: blood flow (QB): 400mL/min; gas flow (QG):7L/min — Abylcap settings
Device: Abylcap® System: blood flow (QB): 400mL/min; gas flow (QG):1.5L/min — Abylcap settings
Device: Abylcap® System: blood flow (QB): 400mL/min; gas flow (QG):3L/min — Abylcap settings
Device: Abylcap® System: blood flow (QB): 400mL/min; gas flow (QG):6L/min — Abylcap settings
Device: Abylcap® System: blood flow (QB): 400mL/min; gas flow (QG):8L/min — Abylcap settings

SUMMARY:
This prospective study includes 5 patients with ARDS (Acute Respiratory Distress Syndrome) treated by mechanical ventilation. In case of respiratory acidosis, extracorporeal CO2 (carbon dioxide)removal might be necessary. We hereby work with the Abylcap system with the oxygenator Lilliput2 as CO2 remover (Bellco, Italy).

The patients (M/V) are older than 18, not pregnant, have a BMI<30, and no contraindication for anticoagulation therapy.

Under standard conditions patients are treated with a blood flow of QB=300mL/min and a gas flow (100% 02) of QG=7L/min. Blood sampling is performed from the arterial bloodline in the patients at 0, 1h, 3h, 24h, 48h, 72h, 96h, and 120h.

A parameter study is also performed to optimise CO2 removal. Herewith, blood samples (1mL) are taken from the inlet and outlet line of the Lilliput2 at the previously mentioned time points and for different flow setting: Blood flow (QB) 200-300-400mL/min and gas flow (QG) 1.5, 3, 6, 7, 8L/min

Blood samples are analysed for the different blood gases from which the extraction in the CO2 remover can be calculated for each setting of QB (blood flow) and QG (gas flow).

ELIGIBILITY:
Inclusion Criteria:

* Patients with ARDS and respiratory acidosis on the intensive care unit
* Treated with the Abylcap system (Bellco, Italy)
* Not pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-02-20 (Actual); Primary Completion 2014-06-13 (Actual); Study Completion 2014-09-12 (Actual)

PRIMARY OUTCOMES:
calculation of CO2 extraction in blood samples during mechanical ventilation | during mechanical ventilation with CO2 removal (max up to 120h)
  Extraction is calculated from the relative difference in blood gases at the inlet and outlet of the CO2 remover.

SECONDARY OUTCOMES:
Based on the extraction rates, the optimum parameter settings are derived | During mechanical ventilation with CO2 removal (max up to 120h)
  Extraction is calculated from the relative difference in blood gases at the inlet and outlet of the CO2 remover.

CONTACTS AND LOCATIONS:
Overall Officials: Sunny Eloot, PhD, MScBME, MScCivE, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Oost-Vlaanderen, Belgium